CLINICAL TRIAL: NCT06296732
Title: Abdominal Neuroblastoma Laparoscopic Surgery Risk Factors Stratification
Acronym: ANLAP-R
Status: Recruiting | Type: Observational
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Collaborators: University Medical Center, Kazakhstan (Other)
Responsible Party: Sponsor
Other Study IDs: NCPHOI-2024-01
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-02

CONDITIONS: Neuroblastoma; Ganglioneuroma; Ganglioneuroblastoma
Keywords: Neuroblastoma; Ganglioneuroma; Ganglioneuroblastoma; Laparoscopic surgery; Minimally-Invasive surgery; IDRF - image-defined risk factors; Risk factors; Difficulty scoring system; Complete resection
MeSH Terms: conditions — Neuroblastoma; Ganglioneuroma; Ganglioneuroblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Duration of surgery intervention — Intraoperative- duration from the beginning of the skin incision to skin suture (min)

SUMMARY:
Surgery plays significant role in treatment of neurogenic tumors, both for benign ganglioneuroma and for high risk neuroblastoma. The world literature has accumulated large experience in laparoscopic surgery for abdominal neuroblastoma. The presence of IDRF (image-defined risk factors) and tumor size (>4-7 cm) are considered as common contraindications for minimally invasive surgery in neuroblastoma. However, the recent studies have shown that presence of IDRF is not an absolute contraindication for laparoscopic surgery. This open-label, nonrandomized, observational, phase III evaluates role and weight of different surgical risk factors (including IDRF, tumor size, tumor localization, tumor volume/patient height ratio, previous open surgical procedures, previous chemotherapy etc.) in the laparoscopic neuroblastoma resections. The aim of this study is to create novel risk factors scoring system for laparoscopic surgery in abdominal neuroblastoma.

DETAILED DESCRIPTION:
After signing informed consent and surgical risk factors assessment (see Study Documents), eligible patients received surgical treatment - laparoscopic neuroblastoma resection. Parameters to be assessed are: duration of surgery intervention, intraoperative complications, blood loss volume, cases and volume of blood transfusion, conversion from laparoscopic to cavity access, surgeon's visual assessment completeness of the tumor resection. During 5 postoperative days patients undergo contrast-enhanced abdominal computed tomography (CT) to control completeness of the tumor resection assessment. Postoperative complications during 30 postoperative days to be accessed. In follow up period 1-, 3- and 5 years local recurrence-free survival to be accessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with neurogenic tumors meeting the criteria of groups I-III:

   Group I
   * low or moderate risk group according to pilot difficulty scoring system (less than 5 points, see supplementary material);
   * no IDRF;

   Group II:
   * low or moderate risk group according to pilot difficulty scoring system (less than 5 points);
   * patients with any number of IDRFs and without central tumor location and/or tumor extension across the midline and/or tumor volume (cm3)/patient height (m) ratio = 28 or more.

   Group III:
   * 2 and more IDRF + central tumor location and/or tumor extension across the midline;
   * 2 and more IDRF + tumor volume (cm3)/patient height (m) ratio = 28 or more;
   * 2 and more IDRF + 2 and more other risk factors according to pilot difficulty scoring system;
   * 1 IDRF + tumor extension across the midline + tumor volume (cm3)/patient height (m) ratio = 28 or more.
2. Age from 0 to 18 years.
3. Preoperative imaging (abdominal contrast-enhanced computed tomography (CT), performed no later than 14 days before the planned surgery).
4. Indications for surgery based on the decision of multidisciplinary experts board in centers- participants.
5. Written voluntary informed consent of the patient and / or his legal representative.

Exclusion Criteria:

1. 3 and more IDRF + central tumor location and/or tumor extension across the midline and/or tumor volume (cm3)/patient height (m) ratio = 28 or more.
2. Severe concomitant pathology, increasing anesthesiologic and surgical risks, via the desicion of the research physician or conclusion by multidisciplinary team in centers- participants.
3. Tumor volume does not technically allow to provide minimally-invasive surgery, based on the conclusion of multidisciplinary experts board team in centers- participants.
4. Therapy strategy: observation

   -

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with abdominal neurogenic tumors in 0-18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-10-26 (Estimated); Study Completion 2031-11-01 (Estimated)

PRIMARY OUTCOMES:
Duration of surgery intervention | Intraoperative
  Pilot difficulty scoring system for laparoscopic surgery in abdominal neuroblastoma

SECONDARY OUTCOMES:
The influence of surgical risk factors | Intraoperative and 30 days postoperative
  The influence of surgical risk factors (see supplementary material) on the surgery results (see supplementary material) and the course of the postoperative period.
Cases of conversion from laparoscopic to cavity access | Intraoperative
Comparison of surgeon's visual assessment of the tumor resection | 5 days postoperative
  Comparison of surgeon's visual assessment of the tumor resection completeness with data from abdominal contrast-enhanced CT, performed in the first 5 days after surgery.
1-, 3-, 5-years local recurrence-free survival | up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of Pediatric Hematology, Oncology and Immunology, Moscow, Russia